CLINICAL TRIAL: NCT03042169
Title: Surgical Resection Plus Chemotherapy Versus Chemotherapy Alone in Oligometastatic Stage IV Gastric Cancer - a Multicenter, Prospective, Open-labeled, Two-armed, Randomized, Controlled Phase III Trial
Brief Title: Surgical Resection Plus Chemotherapy Versus Chemotherapy Alone in Oligometastatic Stage IV Gastric Cancer
Acronym: SURGIGAST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: default inclusion
Sponsor: University Hospital, Lille (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015_07; 2016-A01265-46 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-01-31; First posted 2017-02-03 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Gastric Adenocarcinoma
Keywords: Stage IV gastric cancer; palliative surgery; chemotherapy; survival; quality of life
MeSH Terms: conditions — Stomach Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continuation of chemotherapy (Active Comparator): Patients assigned to arm A will continue to receive the same chemotherapy regimen they received before randomization. Chemotherapy should be restarted between D1 and D30 after randomization.
  In case of poor tolerance to the induction chemotherapy, alternative chemotherapy regimen might be discussed, according to local standards and national guidelines (www.tncd.org).
  Interventions: Drug: Preoperative Chemotherapy; Drug: Postoperative chemotherapy
- surgical removal of the primary tumour and treatment of the metastatic site followed by chemotherapy (Experimental): Patients assigned to arm B will undergo gastrectomy (subtotal or total according to the location of the primary tumour) between D1 and D30 after randomization.
  Subtotal gastrectomy is recommended if it allows a complete resection of the primary tumour to limit postoperative morbidity in such metastatic situations, based on the results of REGATTA
  Interventions: Procedure: Surgery; Drug: Postoperative chemotherapy

INTERVENTIONS:
Drug: Preoperative Chemotherapy — Standard chemotherapy regiments according to risk of recurrence
  Arms: continuation of chemotherapy
Procedure: Surgery — the surgical treatment will undergo gastrectomy between D1 and D30 after randomization.
  Other Names: surgical removal of the primary tumour followed by chemotherapy
  Arms: surgical removal of the primary tumour and treatment of the metastatic site followed by chemotherapy
Drug: Postoperative chemotherapy — Chemotherapy should be restarted between D1 and D30 post-randomization

SUMMARY:
Surgical resection of the primary tumour and treatment of the metastatic site in oligometastatic stage IV metastatic gastric adenocarcinoma enhances survival and improves quality of life with acceptable postoperative morbidity and mortality in a selected group of operable patients with only one metastatic site that does not progress under chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis of UICC stage IV gastric adenocarcinoma with histological proof of the primary tumour (with HER2 status, PCC histology and MMR status available and SRC histology available on anatomo-pathology reports)
2. Without any form of previous treatment (surgery and / or chemotherapy and / or radiotherapy) for this diagnosis other than local endoscopic treatment. Note : 3. pPatients having received first line chemotherapy for at least 2 months and completing inclusion/exclusion criteria can be included in the study at V2
3. Locally resectable primary tumour and oligometastatic lesion accessible to surgical resection or local ablation procedure
4. Oligometastatic lesion : Retro-Peritoneal Lymph Node Metastases (RPLM) and/or another metastatic lesion on only one organ (solid organ, lymph node or limited localised peritoneal carcinomatosis with PCI < 7) according to the following non-exhaustive list of definitions:

   1. RPLM: para-aortal, intra-aorto-caval, para-pancreatic or mesenteric lymph node(s). Note: in duodenum invading gastric cancer, retro-pancreatic nodes are not regarded as metastatic sites
   2. Other acceptable limited metastatic lesions:

      * Localized potentially operable peritoneal carcinomatosis: PCI < 7 including uni or bilateral Krukenberg tumors (ovarian metastases)
      * Liver: maximum of 5 metastatic lesions that are potentially resectable
      * Lung: unilateral involvement, potentially resectable
      * Uni- or bilateral adrenal gland metastases
      * Extra-abdominal lymph node metastases such as supraclavicular or cervical lymph node involvement
      * Localized bone involvement (defined as being within one radiation field) Notes: 1. Patients with more than one metastatic site in only one organ are eligible. 2. In case of doubt for considering whether a metastatic site is limited or not, please submit the case with relevant anonymised information to the medical coordinator of the study for approval. 6. Only one solid organ metastatic site (hepatic, lung, adrenal gland, bone, brain...). Patients with more than one metastatic lesion in only one organ are eligible
5. ECOG performance status 0 or 1
6. Man or women aged ≥ 18 years and ≤ 80 years
7. For surgery and/or chemotherapy, adequate cardiac, respiratory, bone marrow, renal and liver functions according to usual practices standards
8. Ability to understand and complete quality of life questionnaires (EORTC QLQ C30 and QLQ STO 22)
9. Negative pregnancy test (urine or serum) performed prior to start the study in for females of childbearing potential with reproductive potential
10. Male and female patients of child-bearing reproductive potential must agree to us an effective method of contraception approved by the investigator during the study and for a minimum of 6 months after the end of study treatment
11. Patient covered by a government Health Insurance
12. Patient who provides a signed written Inform Consent

Exclusion Criteria:

1. Other histological subtype than adenocarcinoma
2. ECOG performance status ≥ 2 2,3 or 4
3. Diffuse peritoneal carcinomatosis (PCI ≥ 7) or significant ascites
4. Metastatic disease involving more than one solid organ metastatic site
5. Primary tumor irresectability and/or metastatic lesion not accessible for resection or local ablation procedure or need for multi-visceral resection with expected high complication rate
6. Contraindication to chemotherapy or surgery according to the multidisciplinary team decision
7. Second uncontrolled malignant tumour
8. Proximal (junctionnal) tumour growth across the Z-line requiring additional trans thoracic oesophageal resectionµ
9. Emergency surgery due to bleeding or perforation
10. Age > 80 years
11. Weight loss ≥ 20% persisting despite appropriate nutritional assistance
12. Severe comorbid conditions that may jeopardize short term outcomes (e.g. cardiac, respiratory, bone marrow, renal or liver insufficiency...)
13. Dihydropyrimidine dehydrogenase Deficiency (DPD)
14. Women who are pregnant or breastfeeding
15. Patients in emergency situations
16. Patients kept in detention and/or under legal protection under psychiatric care and/or interned in a social or psychiatric institution
17. Adult patient under legal protection or in the incapacity to express his/her consent
18. Patient not covered by a health insurance system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Overall survival | Between the date of randomisation to the date of death whatever the cause,assessed up to 2 years

SECONDARY OUTCOMES:
EORTC QLQ C30 | Every 3 months during 2 years
QLQ STO 22 questionnaires | Every 3 months during 2 years
Progression free survival | from randomisation to the date of documented progression according to RECIST or death whatever the cause,assessed up to 2 years
Surgery related postoperative morbidity-mortality | within 30 days and 90 days
  grade III, IV and V and complications according to the Dindo-Clavien classification
Specific complications related to treatment of the metastatic site | within 30 days and 90 days post-treatment
  grade III, IV and V complications according to the Dindo-Clavien classification for surgical treatment strategy and grade III, IV and V adverse reactions according to the NCI-CTCAE v5.0 for other treatment strategies (i.e. HIPEC, radiofrequency, microwave and radiotherapy).
Chemotherapy related toxicities : grade III, IV and V toxicities according to the NCI-CTCAE v5.0 | Every 3 months during 2 years]
Overall cumulative duration of hospitalisation | throughout the duration of the study, during 2 years
  calculated in days from randomization
Number of interventional palliative procedures per patient | throughout the duration of the study, during 2 years
  mean per patient from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Piessen, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Ico - Site Gauducheau - St Herblain, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: No